CLINICAL TRIAL: NCT05337891
Title: Sensitivity of Repetitive Nerve Stimulation Performed in the Evening vs in the Morning and With Single vs Repeated Effort in Myasthenia Gravis
Brief Title: Sensitivity of Repetitive Nerve Stimulation Performed in the Evening vs in the Morning in Myasthenia Gravis
Status: Recruiting | Type: Observational
Sponsor: Jagiellonian University (Other)
Responsible Party: Principal Investigator, Jakub Antczak, Principal Investigator, Jagiellonian University
Other Study IDs: JagiellonianU70
Record Dates: First submitted 2022-04-13; First posted 2022-04-20 (Actual); Last update posted 2024-10-10 (Actual); Status verified 2024-10

CONDITIONS: Myasthenia Gravis
Keywords: Myasthenia Gravis; Repetitive Nerve Stimulation; effort; Morning; Evening
MeSH Terms: conditions — Myasthenia Gravis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with suspected or diagnosed myasthenia gravis: Patients with suspected or diagnosed myasthenia gravis (ocular and generalized form), aged 18-80, both sexes, with performed or planned determination of anti-acetylcholine receptor antibodies and muscle-specific tyrosine kinase antibodies

SUMMARY:
Myasthenia gravis (MG) is the autoimmune disorder affecting the neuromuscular junction, characterized by fatigue, which increases gradually through the day. The repetitive nerve stimulation (RNS) remains the key diagnostic test in MG, however its sensitivity, especially in ocular form of MG is not satisfactory. In this study, investigators want to assess the impact of the time of the day on the sensitivity of the RNS. We hypothesize the RNS performed in the evening may be more sensitive than in the morning.

DETAILED DESCRIPTION:
Myasthenia gravis (MG) is the autoimmune disorder affecting the neuromuscular junction with morbidity estimated at 70-320 per 1 000 000. The main symptom is the fatigue, which increases gradually through the day and also after exercise. The repetitive nerve stimulation (RNS) remains the key diagnostic test. In RNS, the peripheral nerve is electrically stimulated with trains of repetitive pulses at constant (e.g. 3Hz) frequency. The electrical responses associated with contraction of the one of respectively innervated muscles are recorded. While in healthy subject the amplitudes of subsequent responses should be similar, in MG they gradually decrease reflecting the insufficiency of neuromuscular junction and being the electrophysiological correlate of the fatigue. RNS is relatively simple, safe as well as time and cost-effective procedure. However, its sensitivity is not satisfactory. Even when voluntary exercise and other provocative methods are implemented, the sensitivity does not exceed 89% in generalized form of MG (where symptoms affect bulbar, limb and other muscles) and 70% in ocular form (where symptoms are limited to bulbar muscles). In some laboratories the sensitivity of detecting the impaired neuromuscular transmission can be increased with the use of the single fiber electromyography. This method is however not widely available as it requires skilled personnel and dedicated software. It is also not specific for MG. Therefore, research effort is still being done to increase the sensitivity of the RNS. The well-known gradual exacerbation of MG-related fatigue through the day let us to hypothesize, the RNS performed in the evening may be more sensitive than in the morning. The primary objective of this study will be therefore a comparison of RNS sensitivity performed in these both times of the day. Additionally, investigators want to assess if adding the second voluntary effort could be another way of improving the RNS-sensitivity. The maximal voluntary effort of the investigated muscle, lasting between 30 seconds and one minute is typically done in the course of the RNS. Usually, one or several trains of five to ten impulses precede it and also several trains follow it. While prolonging the effort over one minute may cause discomfort or problems with adherence, adding second one-minute effort, separated from the first by several trains should be suitable and well tolerable. It will prolong the whole procedure by approximately six minutes minutes.

Diagnostic procedure: In every recruited patient, RNS will be done thrice at 8:30 a.m., 8:50 a.m. and 2:30 p.m. on the same day or at 8:30 a.m. and 8:50 a.m. on one day and at 2:30 p.m. on the subsequent day. To exclude peripheral neuropathy, before the first RNS, the sensory nerve conduction study will be performed on the sural nerve and the motor conduction study on the tibial nerve on the nondominant side. To exclude myopathy, before the first RNS, the needle electromyography will be performed on the biceps brachii, of dominant side. Also, before the first RNS, the Myasthenia Gravis - Activities of Daily Living Score (MG-ADL) will be filled out. Every RNS will comprise investigation of the nasalis and trapezius muscles on the clinically more affected side or on the nondominant side when lateralization will not be evident. Investigation of every muscle will include two, 3Hz trains of ten supramaximal electric stimuli, separated by 1 minute interval. Then the 1 minute of maximal voluntary effort will follow and after that six 3Hz trains of ten supramaximal stimuli, separated by 1-minute intervals. The first or the second RNS (at 8:30 or at 8:50 a.m.) will include additional 1 minute of maximal voluntary effort, followed by additional six 3Hz trains of ten supramaximal stimuli, separated by 1-minute intervals. The allocation of the additional voluntary effort and subsequent six trains to the first or to the second RNS will be done randomly. The randomization list will be created via the website www.randomization.com using blocks of five subjects. The amplitude drop (the decrement) of the fourth response (out of 10 in every train) >=10% with respect to the first response will be considered abnormal (indicative of impaired neuromuscular transmission). The whole RNS will be considered abnormal (indicative of impaired neuromuscular transmission) when the decrement >=10% will be repeatable in at least several trains in at least one out of two tested muscles. The temperature of the skin will be maintained at 35 Celsius. If being taken, the acetylcholinesterase inhibitors will be withheld 12 hours before the first RNS.

ELIGIBILITY:
Inclusion Criteria:

* Patients with suspected or diagnosed myasthenia gravis (ocular and generalized form)
* Patients with performed or planned determination of anti-AChrR and anti-MUSK antibodies.
* Disease severity of at least 1 in the classification of the severity of myasthenia gravis according to the recommendations of the Myasthenia Gravis Foundation of America

Exclusion Criteria:

* respiratory failure
* severe bulbar symptoms
* pharmacotherapy with substances that may worsen neuromuscular transmission disorders
* current infection
* coexisting diseases of the peripheral nervous system which may affect the result of the fatigue test, e.g. polyneuropathy or myopathy
* cognitive and behavioral disorders that may negatively affect patient's adherence to study protocol
* Medication with steroids due to myasthenia
* Severity of myasthenia that makes the discontinuation of acetylcholinesterase inhibitors unsafe.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Convenience sample of 40 people with suspected or diagnosed myasthenia gravis (ocular and generalized form). Patients will be recruited from the Outpatient Clinic of the Neurology Clinic of University Hospital in Cracow
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2022-06-03 (Actual); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Difference in the highest decrement between investigation of nasalis during morning and evening RNS | Through study completion, an average of 1 year.
  Difference in the highest decrement between investigation of nasalis during morning (at 8:30 or 8:50 a.m.) RNS with single one-minute voluntary effort and RNS at 2:30 p.m.
Difference in the highest decrement between investigation of trapezius during morning and evening RNS | Through study completion, an average of 1 year.
  Difference in the highest decrement between investigation of trapezius during morning (at 8:30 or 8:50 a.m.) RNS with single one-minute voluntary effort and RNS at 2:30 p.m.
Difference in the highest decrement between investigation of nasalis during morning RNS with single and with two voluntary efforts | Through study completion, an average of 1 year.
  Difference in the highest decrement between investigation of nasalis during morning (at 8:30 or 8:50 a.m.) RNS with single one-minute voluntary effort and RNS with two one-minute voluntary efforts.
Difference in the highest decrement between investigation of trapezius during morning RNS with single and with two voluntary efforts | Through study completion, an average of 1 year.
  Difference in the highest decrement between investigation of trapezius during morning (at 8:30 or 8:50 a.m.) RNS with single one-minute voluntary effort and RNS with two one-minute voluntary efforts.

SECONDARY OUTCOMES:
Difference in the percentage of abnormal RNS results between RNS performed in the morning and in the evening | Through study completion, an average of 1 year.
  Difference in the percentage of abnormal RNS results between RNS with single one-minute voluntary effort performed in the morning (at 8:30 or 8:50 a.m.) and RNS performed at 2:30 p.m.
Difference in the percentage of abnormal RNS results between RNS performed in the morning with single and with two voluntary efforts | Through study completion, an average of 1 year.
  Difference in the percentage of abnormal RNS results between RNS with single one-minute voluntary effort performed at 8:30 or 8:50 a.m. and RNS with two one-minute voluntary efforts.
Correlation between the highest decrement during morning RNS with single one-minute voluntary effort and the MG-ADL score | Through study completion, an average of 1 year.
  Correlation between the highest decrement during RNS with single one-minute voluntary effort, performed at 8:30 or 8:50 AM and the MG-ADL score
Correlation between the highest decrement during RNS with two one-minute voluntary efforts and the MG-ADL score | Through study completion, an average of 1 year.
  Correlation between the highest decrement during RNS with two one-minute voluntary efforts, and the MG-ADL score
Correlation between the highest decrement during evening RNS and the MG-ADL score | Through study completion, an average of 1 year.
  Correlation between the highest decrement during RNS performed at 2:30 p.m. and the MG-ADL score

CONTACTS AND LOCATIONS:
Overall Officials: Jakub M Antczak, MD, Principal Investigator — Jagiellonian University Medical College, Department of Neurology
Locations (1):
- Jagiellonian University Medical College, Department of Neurology, Krakow, Lesser Poland Voivodeship, Poland

IPD SHARING:
Plan to Share IPD: Yes
After completing the study, the age and gender of participants as well as the scores and results of all outcome measurements together with electrophysiological recordings will be made available to other researchers on request.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: The data will become available after the study results will be published.
Access Criteria: On request sent by e-mail to jakub.antczak@uj.edu.pl

REFERENCES:
- [Result] Witoonpanich R, Dejthevaporn C, Sriphrapradang A, Pulkes T. Electrophysiological and immunological study in myasthenia gravis: diagnostic sensitivity and correlation. Clin Neurophysiol. 2011 Sep;122(9):1873-7. doi: 10.1016/j.clinph.2011.02.026. Epub 2011 Mar 17. PMID 21419697
- [Result] Bou Ali H, Salort-Campana E, Grapperon AM, Gallard J, Franques J, Sevy A, Delmont E, Verschueren A, Pouget J, Attarian S. New strategy for improving the diagnostic sensitivity of repetitive nerve stimulation in myasthenia gravis. Muscle Nerve. 2017 Apr;55(4):532-538. doi: 10.1002/mus.25374. Epub 2017 Jan 3. PMID 27511866
- [Result] Wolfe GI, Herbelin L, Nations SP, Foster B, Bryan WW, Barohn RJ. Myasthenia gravis activities of daily living profile. Neurology. 1999 Apr 22;52(7):1487-9. doi: 10.1212/wnl.52.7.1487. PMID 10227640
- [Result] Jaretzki A 3rd, Barohn RJ, Ernstoff RM, Kaminski HJ, Keesey JC, Penn AS, Sanders DB. Myasthenia gravis: recommendations for clinical research standards. Task Force of the Medical Scientific Advisory Board of the Myasthenia Gravis Foundation of America. Neurology. 2000 Jul 12;55(1):16-23. doi: 10.1212/wnl.55.1.16. No abstract available. PMID 10891897